CLINICAL TRIAL: NCT05315284
Title: The Clinical and Radiological Outcomes of the Use of Titanium Elastic Nail in The Fixation of Fresh Non-comminuted Fracture Mid-shaft Clavicle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Salah Mohamed, Resident Doctor, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-02-08
Record Dates: First submitted 2022-03-18; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Fracture Clavicle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with fresh non-comminuted fracture mid-shaft clavicle (Other)
  Interventions: Procedure: the Use of Titanium Elastic Nail in The Fixation of Fresh Non-comminuted Fracture Mid-shaft Clavicle

INTERVENTIONS:
Procedure: the Use of Titanium Elastic Nail in The Fixation of Fresh Non-comminuted Fracture Mid-shaft Clavicle — Fixation of Fresh Non-comminuted Fracture Mid-shaft Clavicle

SUMMARY:
The Clinical and Radiological Outcomes of the Use of Titanium Elastic Nail in The Fixation of Fresh Non-comminuted Fracture Mid-shaft Clavicle

DETAILED DESCRIPTION:
Introduction:

The midshaft clavicle fractures account for 3 to 5% of all injuries and 70 to 80% of all clavicle fractures.[1,2] In young adults, these fractures are usually related to sports or vehicle accidents, whereas in children and elderly, they are usually related to falls.[1,2] In general, clavicle fractures are treated conservatively and have a good outcome. In 1960, Neer reported a non-union rate of 0.1% with conservative treatment[3] and Rowe corroborated these findings in 1968 and showed a nonunion rate of 0.8% in conservatively managed patients.[4] Since then, however, other authors have failed to demonstrate similar good results with conservative treatment.[5,6] This may be due to the fact that the initial series included children and adolescents and their enormous potential for bone healing may have skewed the results, and that patient-based scoring systems were not used in the initial series to record the outcome.[7] Hill et al. showed that displacement of more than 20 mm resulted in 15% non-union and 18% of the patients had thoracic outlet syndrome following union.[5] McKee et al. noted reduced patient satisfaction due to asymmetry and cosmesis following malunion in patients with more than 20 mm shortening.[6] Hence, more recently, there has been a trend toward surgical fixation.

Surgery has been indicated for completely displaced fractures, potential skin perforation, shortening of clavicle by more than 20 mm, neurovascular injury, and floating injury.[8] The gold standard for the surgical treatment has been open reduction and plate fixation through a large incision.[8] Other surgical options include intramedullary pinning with Kirschner wire, Rush pins, Knolwes pin, Steinman pin, Haige pin, ESIN (elastic stable intramedullary nailing), and external fixation.[9] Intramedullary fixation for clavicular fractures was first described by Peroni in 1950.[10] A systematic review showed relative risk reduction of 72% and 57% for non-union when using intramedullary fixation and plate fixation, respectively, when compared with non-operative treatment of midshaft clavicle fractures.[11] Intramedullary devices behave as internal splints that maintain alignment without rigid fixation. The use of an intramedullary device carries advantages of a smaller incision, less soft tissue dissection, load sharing fixation with relative stability that encourages copious callus formation.[12] The titanium ESIN has been successfully used in fixation of pediatric long bone fractures. One advantage of the titanium ESIN is that it can block itself in the bone and provide a three-point fixation within the Sshaped clavicle.[8,13] However, some studies have shown a relatively high complication rate and technical difficulties with intramedullary nailing.[7,8] The aim of this study was to investigate the union rate and complication rate of our patients with displaced midshaft clavicle fractures treated with titanium ESIN. Aim of the study Investigating the union rate and complications rate following titanium elastic stable intramedullary nailing (ESIN) for midshaft non-comminuted clavicle fractures with >20 mm shortening/displacement. Materials and methods Place of the study: Orthopaedics and Traumatology Department, Sohag University Hospital. Type of the study: Prospective study. Study period: from December,2021 till December,2022. Inclusion criteria: (1) Type IIA2 (angulation > 45 ) or IIB1 (shortening or overlapping displacement length > 2 cm) fresh unilateral midshaft clavicular fractures according to Robinson classification. (2) Patient without underlying diseases such as primary hypertension and cardiac diseases. Exclusion criteria: (1) pathological fractures. (2) multiple injuries of upper limbs. (3) open fractures. (4) combined with injuries of blood vessels or nerves. (5) other diseases which affected the functions of upper limbs. (6) Proximal and distal clavicular fractures. (7) Comminuted clavicular fractures. Preoperative assessment: (1) Clinical evaluation: pain, tenderness, deformity, shortening, skin tethering and loss of function. (2) Radiological assessment: plain X-ray imaging is the corner stone for establishing the diagnoses of clavicular fractures. CT scans can be used to exclude comminuted clavicular fractures if the comminution of the fracture couldn't be visualized by the plain X-ray studies (3) Laboratory assessment: routine laboratory investigations for any surgery.

Standard protocol approvals and patient consents:

This study will be approved by the Medical Research Ethics committee at faculty of medicine, Sohag University. An informed written consent will be obtained from each patient.

Surgical technique:

After administration of anesthesia, the patient is placed in beach chair position with injured extremity prepared and draped from the midline to the upper arm. Care is taken to make sure that the sternoclavicular joint was accessible for the entry point. Preoperatively, the shoulder region is screened using image intensifier to confirm this access. A vertical skin incision is made just lateral to the sternoclavicular joint. The subcutaneous fat is incised along with platysma. The pectoral fascia is divided in line with the skin incision followed by careful elevation of the underlying musculature from the clavicle. The entry point in the anterior cortex with a 3.2 mm drill bit and guide. The entry portal may be enlarged with an awl and appropriate sized titanium ESIN is inserted (The size of the nail was measured using this formula = 0.4 × canal diameter in mm). Attempt is made to close reduce the fracture. If the fracture could not be reduced by closed means, then a separate vertical incision is used at the fracture site to aid fracture reduction. Vertical incision is used as it is parallel to Langer's lines and minimizes the risk of damage to supraclavicular nerves to avoid dysesthesia of skin and scar neuromas. The nail is used to create a path in the lateral end of the clavicle for subsequent easy access.

The nail is then passed from the medial side and across the reduced fracture into the lateral end of clavicle.

Postoperative management:

All patients are treated with arm sling after operation for 6 weeks. In addition, 3 days after surgery, patients are allowed to do passive anteflexion and abduction motion of shoulder joint under the guidance of physiotherapists, and the motion range could be increased gradually depending on the degree of pain. However, the range of passive anteflexion and abduction motion is kept within 90 degrees in 6 weeks after surgery, and the weight-bearing exercise is not allowed. The range of passive and active motion is increased gradually according to the condition of fracture union and the weight-bearing exercise is started gradually after 6 weeks post-operatively. The postoperative follow-up visits are scheduled every two weeks until bone union and every 3 months after bone union. Post-Operative Evaluation

Evaluation of therapeutic efficiency:

The operative data is recorded and analyzed, including operation time, blood loss, hospital stays and postoperative complications. The standards of bone union includes the formation of continuous callus and the disappearance of fracture line, no tenderness of the fracture ends, and no subjective pain when performing active sports and weight-bearing activities on the clinical examinations.

Scoring system:

Improvement of subjective pain is assessed using a visual analog scale (VAS) at 1 day before surgery and 3 days after surgery. The flexion and abduction motion ranges of shoulder joint were recorded from one day before surgery to the last follow-up.24 Shoulder function is assessed with the Constant-Murley score (range: 0-100 points, best: 100) and the Disabilities of the Arm, Shoulder and Hand (DASH) score (range: 0- 100 points, best: 0) at the last follow-up. In detail, Constant-Murley scores are categorized as follows: excellent (90-100), good (80-89), satisfactory (70-79), and fair (<70). DASH scores of 0-10 are considered as an excellent result, and score >40 is associated with poor shoulder function.

ELIGIBILITY:
Inclusion Criteria:

* : (1) Type IIA2 (angulation > 45 ) or IIB1 (shortening or overlapping displacement length > 2 cm) fresh unilateral midshaft clavicular fractures according to Robinson classification. (2) Patient without underlying diseases such as primary hypertension and cardiac diseases.

Exclusion Criteria:

* (1) pathological fractures. (2) multiple injuries of upper limbs. (3) open fractures. (4) combined with injuries of blood vessels or nerves. (5) other diseases which affected the functions of upper limbs. (6) Proximal and distal clavicular fractures. (7) Comminuted clavicular fractures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The Clinical Outcome of the Use of Titanium Elastic Nail in The Fixation of Fresh Non-comminuted Fracture Mid-shaft Clavicle | 3 months
  Investigating the union rate and complications rate following titanium elastic stable intramedullary nailing (ESIN) clinically for midshaft non-comminuted clavicle fractures with >20 mm shortening/displacement.
The Radiological Outcome of the Use of Titanium Elastic Nail in The Fixation of Fresh Non-comminuted Fracture Mid-shaft Clavicle | 3 months
  Investigating the union rate and complications rate following titanium elastic stable intramedullary nailing (ESIN) radiologically for midshaft non-comminuted clavicle fractures with >20 mm shortening/displacement.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. Duan X, Zhong G, Cen S, Huang F, Xiang Z. Plating versus intramedullary pin or conservative treatment for midshaft fracture of clavicle: A meta-analysis of randomized controlled trials. J Shoulder Elbow Surg 2011;20:1008-15. 2. Schiffer G, Faymonville C, Skouras E, Andermahr J, Jubel A. Midclavicular fracture: not just a trivial injury: Current treatment options. Dtsch Arztebl Int 2010;107:711-7. 3. Neer CS 2nd. Nonunion of the clavicle. J Am Med Assoc 1960;172:1006-11. 4. Rowe CR. An atlas of anatomy and treatment of midclavicular fractures. Clin Orthop Relat Res 1968;58:29-42. 5. Hill JM, McGuire MH, Crosby LA. Closed treatment of displaced middle-third fractures of the clavicle gives poor results. J Bone Joint Surg Br 1997;79:537-9. 6. McKee MD, Pedersen EM, Jones C, Stephen DJ, Kreder HJ, Schemitsch EH. Deficits following nonoperative treatment of displaced midshaft clavicular fractures. J Bone Joint Surg Am 2006;88:35-40. 7. Smekal V, Irenberger A, Struve P, Wambacher M, Krappinger D, Kralinger FS. Elastic stable intramedullary nailing versus nonoperative treatment of displaced midshaft clavicular fractures-a randomized, controlled, clinical trial. J Orthop Trauma 2009;23:106-12. 8. Frigg A, Rillmann P, Perren T, Gerber M, Ryf C. Intramedullary nailing of clavicular midshaft fractures with the titanium elastic nail: Problems and complications. Am J Sports Med 2009;37:352-9. 9. Khalil A. Intramedullary screw fixation for midshaft fractures of the clavicle. Int Orthop 2009;33:1421-4. 10. Peroni L. Medullary osteosynthesis in the treatment of clavicle fractures. Arch Ortop 1950;63:398-405. 11. Zlowodzki M, Zelle BA, Cole PA, Jeray K, McKee MD, EvidenceBased Orthopaedic Trauma Working G. Treatment of acute midshaft clavicle fractures: Systematic review of 2144 fractures: on behalf of the Evidence-Based Orthopaedic Trauma Working Group. J Orthop Trauma 2005;19:504-7. 12. Millett PJ, Hurst JM, Horan MP, Hawkins RJ. Complications of clavicle fractures treated with intramedullary fixation. J Shoulder Elbow Surg 2011;20:86-91. 13. Mueller M, Rangger C, Striepens N, Burger C. Minimally invasive intramedullary nailing of midshaft clavicular fractures using titanium elastic nails. J Trauma 2008;64:1528-34. 14. Dawson J, Hill G, Fitzpatrick R, Carr A. The benefits of using patient-based methods of assessment. Medium-term results of an observational study of shoulder surgery. J Bone Joint Surg Br 2001;83:877-82. 15. Beaton DE, Wright JG, Katz JN, Upper Extremity Collaborative G. Development of the QuickDASH: Comparison of three itemreduction approaches. J Bone Joint Surg Am 2005;87:1038-46. 16. Canadian Orthopaedic Trauma S. Nonoperative treatment compared with plate fixation of displaced midshaft clavicular fractures. A multicenter, randomized clinical trial. J Bone Joint Surg Am 2007;89:1-10. 17. Mullaji AB, Jupiter JB. Low-contact dynamic compression plating of the clavicle. Injury 1994;25:41-5. 18. Schuind F, Pay-Pay E, Andrianne Y, Donkerwolcke M, Rasquin C, Burny F. External fixation of the clavicle for fracture or nonunion in adults. J Bone Joint Surg Am 1988;70:692-5. 19. Ferran NA, Hodgson P, Vannet N, Williams R, Evans RO. Locked intramedullary fixation vs plating for displaced and shortened mid-shaft clavicle fractures: A randomized clinical trial. J Shoulder Elbow Surg 2010;19:783-9. 20. Kleweno CP, Jawa A, Wells JH, O'Brien TG, Higgins LD, Harris MB. Midshaft clavicular fractures: Comparison of intramedullary pin and plate fixation. J Shoulder Elbow Surg 2011;20:1114-7. 21. Liu HH, Chang CH, Chia WT, Chen CH, Tarng YW, Wong CY. Comparison of plates versus intramedullary nails for fixation of displaced midshaft clavicular fractures. J Trauma 2010;69:E82-7. 22. Smekal V, Irenberger A, Attal RE, Oberladstaetter J, Krappinger D, Kralinger F. Elastic stable intramedullary nailing is best for midshaft clavicular fractures without comminution: Results in 60 patients. Injury 2011;42:324-9. 23. Jubel A, Andemahr J, Bergmann H, Prokop A, Rehm KE. Elastic stable intramedullary nailing of midclavicular fractures in athletes. Br J Sports Med 2003;37:480-3; discussion 4. 24. Chen YF, Wei HF, Zhang C, Zeng BF, Zhang CQ, Xue JF. Retrospective comparison of titanium elastic nail (TEN) and reconstruction plate repair of displaced midshaft clavicular fractures. J Shoulder Elbow Surg 2012;21:495-501. 25. Smekal V, Oberladstaetter J, Struve P, Krappinger D. Shaft fractures of the clavicle: Current concepts. Arch Orthop Trauma Surg 2009;129:807-15.